CLINICAL TRIAL: NCT02084212
Title: Study of Retinal Sensitivity by Microperimetry During Epiretinal Membrane Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: ISAICO-MUSELIER AOI 2011
Record Dates: First submitted 2014-03-05; First posted 2014-03-11 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Epiretinal Membrane Surgery

ARMS (1):
- Patients about to undergo epiretinal membrane surgery (Other)
  Interventions: Other: Microperimetry

INTERVENTIONS:
Other: Microperimetry

SUMMARY:
The aim of this research is to assess current care by studying macular function using microperimetry and by then comparing visual acuity results with OCT (Optical Coherence Tomography) data.

The examinations performed are those usually done in the follow-up of epiretinal membrane surgery, apart from microperimetry which is an examination of the central visual field. Patients who undergo ERM surgery usually have a follow-up examination at 1 month, 3 months and 6 months after the surgery. The consultation includes an assessment of visual acuity, a fundus examination an SD-OCT of the retina. The present protocol will require no additional visits. The microperimetry will be done in addition to the usual follow-up examinations after ERM surgery.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided consent,
* Patients about to undergo idiopathic epiretinal membrane surgery,
* Patients undergoing first-line macular surgery

Exclusion Criteria:

* Persons not covered by national health insurance
* Preexisting disease of macula/epiretinal membrane (ARMD, chorioretinal scarring)
* Preoperative amblyopic eye
* Insufficiently transparent media making it impossible to do the examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2015-04-24 (Actual); Study Completion 2015-04-24 (Actual)

PRIMARY OUTCOMES:
Change of visual acuity in ETDRS (Early Treatment Diabetic Retinopathy Study) scale | Up to 6 months after the operation.
Anomalies observed in the outer layers of retina | Up to 6 months after the operation
Evaluation of retinal sensitivity by microperimetry | Up to 6 months after the operation

SECONDARY OUTCOMES:
Abnormal surface autofluorescence | Up to 6 months after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France